CLINICAL TRIAL: NCT03611608
Title: A Phase 1 Randomized, Placebo-Controlled Study to Determine the Effect of LY3316531 on Capsaicin-Induced Dermal Blood Flow in Healthy Male Subjects
Brief Title: A Study of LY3316531 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 16667; I9H-MC-FFAB (Other: Eli Lilly and Company); 2018-000710-38 (EudraCT Number)
Record Dates: First submitted 2018-07-27; First posted 2018-08-02 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- 300 mg LY3316531 Dose 1 (Experimental): LY3316531 administered IV
  Interventions: Drug: LY3316531
- LY3316531 Dose 2 (Experimental): The optional additional cohort (Dose 2) was not implemented as the data desired for treatment effect on dermal blood flow (DBF) was generated at the initial Dose 1 (300mg LY3316531)
  LY3316531 administered IV
  Interventions: Drug: LY3316531
- Placebo (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3316531 — Administered IV
  Arms: 300 mg LY3316531 Dose 1; LY3316531 Dose 2
Drug: Placebo — Administered IV
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess study drug activity by giving LY3316531 or placebo into a vein in the arm and then measuring blood flow of the skin, after capsaicin is applied to skin's surface. The study will last about 16 weeks inclusive of the screening period.

ELIGIBILITY:
Inclusion Criteria:

* Must be healthy males
* Must be abstinent or use condoms with spermicide as well as 1 additional highly effective method of contraception or effective method of contraception during the study and for 5 months following dosing of study drug
* Must have a body mass index between 18 to 32.0 kilogram per meter square (kg/m²), inclusive, and a minimum body weight of 50 kilogram (kg)
* Must have suitable skin characteristics for the dermal capsaicin challenge and have demonstrated at least a 100 percent (%) increase in dermal flow following capsaicin challenge as part of the screening procedures and measured through laser Doppler imaging (LDI)

Exclusion Criteria:

* Must not have evidence of clinically significant active infection, fever of 100.5 degrees Fahrenheit (°F) (38 degrees Centigrade (°C)) or above, at baseline
* Must not show evidence of active or latent tuberculosis (TB)
* Must not have received live, attenuated live, or non-live vaccine(s) within 28 days of screening or intend to receive during the study
* Must not be immunocompromised
* Must not have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Must not have significant allergies to humanised monoclonal antibodies
* Have a history of multiple or severe allergies or has had an anaphylactic reaction to prescription or nonprescription drugs or food
* Must not have had any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin
* Must not have eczema, scleroderma, psoriasis, dermatitis, keloids, tumors, ulcers, burns, flaps, or grafts on their forearm or other abnormality of the skin that may interfere with the study assessments
* Must avoid excess tanning throughout the study and cannot cover forearms for 24 hours prior to each treatment period
* Must not have excessive hair growth on the volar surface of the forearm or currently using lotions, oils, depilatory preparations, or other topical treatments on a regular basis that cannot be discontinued for the duration of the study; participant must not have used any topical treatments within 7 days of the start of the study

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri, 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician., Leuven, Belgium

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received placebo as a single saline intravenous (IV) infusion.
  Capsaicin-induced Dermal Blood Flow (DBF): Topical doses of 20 microliter (µL) capsaicin (1000 microgram (µg)/20 µL) applied to 2 different locations on the participant's forearm to induce an increase in dermal blood flow. A 20 µL topical dose of vehicle was applied to a third location on the forearm.
- 300 Milligram (mg) LY3316531: Participants received a single 300 milligram (mg) LY3316531 IV infusion.
  Capsaicin-induced DBF: Topical doses of 20 microliter (µL) capsaicin [1000 microgram (µg)/20 microliter (µL)] applied to 2 different locations on the participant's forearm to induce an increase in dermal blood flow. A 20 µL topical dose of vehicle was applied to a third location on the forearm.
Period: Overall Study
Arm/Group | Placebo | 300 Milligram (mg) LY3316531
Started | 4 | 12
Received at Least One Dose/Injection | 4 | 12
Completed | 4 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received at least one injection of LY3316531 or Placebo.
Groups:
- Placebo: Participants received placebo as a single saline IV infusion.
  Capsaicin-induced DBF: Topical doses of 20 microliter (µL) capsaicin [1000 microgram (µg)/20 microliter (µL)] applied to 2 different locations on the participant's forearm to induce an increase in dermal blood flow. A 20 µL topical dose of vehicle was applied to a third location on the forearm.
- 300 mg LY3316531: Participants received a single 300 mg LY3316531 IV infusion.
  Capsaicin-induced DBF: Topical doses of 20 microliter (µL) capsaicin (1000 microgram (µg)/20 µL) applied to 2 different locations on the participant's forearm to induce an increase in dermal blood flow. A 20 µL topical dose of vehicle was applied to a third location on the forearm.
- Total: Total of all reporting groups
Arm/Group | Placebo | 300 mg LY3316531 | Total
Number analyzed (Participants) | 4 | 12 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.0 (7.7) | 26.6 (8.5) | 30.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 4 | 12 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 12 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 4 | 12 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 4 | 12 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Capsaicin-Induced Dermal Blood Flow Following LY3316531 Compared to Placebo
Description: To assess target neutralization of calcitonin gene-related peptide by LY3316531 versus placebo, the capsaicin-induced dermal blood flow was measured at baseline (before administration of LY3316531 or placebo) as well as 24 days after a single intravenous dose of LY3316531 or placebo
Time Frame: Baseline, Day 24
Population: All participants who received at least one injection of LY3316531 or Placebo.
Measure: Mean (Standard Deviation); unit: milliliter/100gram/minute (mL/100g/min)
Groups:
- Placebo: Participants received placebo as a single saline IV infusion.
  Capsaicin-induced DBF: Topical doses of 20 microliter (µL) capsaicin (1000 microgram (µg)/20 µL) applied to 2 different locations on the participant's forearm to induce an increase in dermal blood flow. A 20 µL topical dose of vehicle was applied to a third location on the forearm.
Arm/Group | Placebo | 300 mg LY3316531
Number analyzed (Participants) | 4 | 12
milliliter/100gram/minute (mL/100g/min) | 327.19 (67.02) | 63.65 (53.31)
Statistical Analysis 1: Comparison: Placebo vs 300 mg LY3316531; Test type: Superiority; p < 0.001, t-test, 1 sided; Mean Difference (Final Values) = 263.54, 90% CI 1-sided [lower limit 207.86]

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3316531
Description: Pharmacokinetics: Maximum Concentration (Cmax) of LY3316531 was reported.
Time Frame: Pre-dose, end of infusion (30min), and 2 hours (h), 6h, 24h, 10 days, 24 days, 38 days, 52 days, 66 days and 80 days post-dose
Population: All participants who received an injection of LY3316531 and contributed PK samples for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (µg/mL)
Arm/Group | 300 mg LY3316531
Number analyzed (Participants) | 12
microgram per milliliter (µg/mL) | 88.2 (15)

3. Secondary Outcome: Pharmacokinetics: Area Under Drug Concentration-Time Curve From Zero to Infinity (AUC[0 ∞]) of LY3316531
Description: Pharmacokinetics: Area Under Drug Concentration-Time Curve From Zero to Infinity (AUC[0 ∞]) of LY3316531 was reported
Time Frame: as for outcome 2
Population: All participants who received an injection of LY3316531 and contributed PK samples for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram*hour per milliliter (µg*h/mL)
Arm/Group | 300 mg LY3316531
Number analyzed (Participants) | 12
microgram*hour per milliliter (µg*h/mL) | 42200 (16)

ADVERSE EVENTS:
Time Frame: Up To 167 days
Description: All participants who received at least one injection of LY3316531 or Placebo.
Arm/Group | Placebo | 300 mg LY3316531
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/12
Other Adverse Events (participants affected / at risk) | 2/4 | 9/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=4) | 300 mg LY3316531 (N=12)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Eyelid skin dryness (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Infusion site reaction (General disorders) | 0 (0) | 1 (1)
Angular cheilitis (Infections and infestations) | 1 (1) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (5)
Pyuria (Infections and infestations) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stress fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Papule (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2019-02-06): https://cdn.clinicaltrials.gov/large-docs/08/NCT03611608/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03611608/SAP_001.pdf